CLINICAL TRIAL: NCT06320639
Title: Driving Simulator and People With Neurocognitive Disorders
Acronym: DRIVS-NCD
Status: Recruiting | Type: Observational
Sponsor: University Gustave Eiffel (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: UGustaveEiffel
Record Dates: First submitted 2024-02-19; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Neurocognitive Disorders
Keywords: Alzheimer's Disease; Vascular encephalopathy; Parkinson's Disease
MeSH Terms: conditions — Neurocognitive Disorders; Alzheimer Disease; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ageing of the population is leading to an increasing number of older drivers on the roads. At the same time, the proportion of older people with pathological ageing and neurocognitive disorders (NCD) is increasing. In terms of road safety, this raises the question of whether these drivers should continue to drive or not. People with NCDs may not be aware of the presence, extent and progression of their cognitive impairment and the impact it can have on daily life, including driving.

Despite their loss of autonomy and medical advice, 22% of people with major NCD continue to drive. In addition, the presence of minor NCD also puts people at a higher risk of road accidents.

However, several studies demonstrated that an NCD does not lead to a systematic and immediate impairment of driving ability and abruptly stopping driving leads to health problems, such as the risk of depression and greatly reduces quality of life.

It is therefore relevant to focus research on driving with people with NCD in order to have a reliable indicator of the person's abilities and the impact of their cognitive impairment on driving activity. The proposed study seeks to meet this need by studying the performance of people with NCD on a driving station (mini-simulator) while assessing their ability to evaluate their performance.

To achieve this goal, people with NCDs will perform tasks on a driving simulator. In addition, after each task on the driving simulator, they will answer questions about how they evaluate their own driving. Two assessors will observe the participants' driving and will estimate their driving performance. By comparing the driver's self-assessment with the assessors' assessment, an "awareness score of driving ability" will be calculated to determine whether the driver correctly assessed his or her performance.

Another project already underway aims to collect similar data from people without a diagnosis of NCDs (control group).

The principal objective of the present study is to compare the driving performance in a simulator and the awareness of driving ability of people with NCDs with those of a control group. Secondary objectives are :

1. to measure driving performance in a simulator and awareness of driving abilities (i.e. self-assessment skills) of people with NCDs.
2. to analyse driving performance and awareness of driving abilities according to the diagnosis and severity of the disorder (i.e. minor or major neurocognitive disorders).
3. to establish a methodology to identify a driver at risk of dangerous driving.

It is mainly an exploratory study however some hypotheses can be made :

* The driving performance and awareness of driving skills of people with NCDs are poorer compared to those of older, control individuals.
* Individuals' driving performance and awareness of driving ability are lower in the presence of major NCDs compared to minor NCDs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Neurocognitive Disorders according to the Diagnostic and Statistical Manual of Mental Disorders-V (DSM-V)
* Normal or corrected vision
* B licence holder with 3+ years driving experience
* Active drivers or drivers who stopped driving less than 2 months ago (time between the medical consultation and the day in the day care hospital)
* For participants able to give consent:

  * Written informed consent to participate in the study
  * Informed consent of the participant in the presence of his/her curator.
* For participants who are not able to receive information and to give consent:

  * Written informed consent of the legal representative (tutor) for participants under tutelage.
  * Signature of a relative (family member and/or trusted person) of the participant
* The participant has to be affiliated to a social security scheme.

Exclusion Criteria:

* History of epilepsy
* People with vestibular disorders, motion sickness or migraines
* Psychiatric history (e.g. schizophrenia)
* Non-stabilized use of antidepressants and/or anxiolytics (started or modified within the last 3 months)
* History of alcoholism
* Use of anti-epileptics
* Osteo-articular pathologies compromising walking

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed with minor or major Neurocognitive Disorders according to the Diagnostic and Statistical Manual of Mental Disorders-V (DSM-V) and recruited from the daycare hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2026-10-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Awareness score of driving ability | Up to 2 hours, from the inclusion until the end of the experiment (2 hours later)
  After each task on the driving simulator, participants answer questions about what they think of their driving performance. Two experimenters write their observations about the participant's performance. Answers are coded in a way that a greater driving performance lead to a greater score.
  The Awareness score is computed by subtracting the score given by the participant to the average of the scores given by the experimenters. The further away from zero the score is, the less aware the participants will be of their abilities. Zero will indicate a perfect assessment of one's abilities.
Driving performance variables measured by the driving simulator | Up to 2 hours, from the inclusion until the end of the experiment (2 hours later)
  For each driving task, the driving variables of interest from the driving simulator will be collected: total braking response time, average speed and lateral lane position for the keeping lane task; distance between vehicles for the car-tracking task; reaction time to unexpected events for the rural and urban driving tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital des Charpennes, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Delphin-Combe F, Coste MH, Bachelet R, Llorens M, Gentil C, Giroux M, Paire-Ficout L, Ranchet M, Krolak-Salmon P. An innovative therapeutic educational program to support older drivers with cognitive disorders: Description of a randomized controlled trial study protocol. Front Neurol. 2022 Jul 18;13:901100. doi: 10.3389/fneur.2022.901100. eCollection 2022. PMID 35923824